CLINICAL TRIAL: NCT05852964
Title: Investigation of Inflammatory and Anti-Inflammatory Gene Expressions in Liver Transplant Patients Before and After the Operation
Brief Title: Inflammatory and Anti-Inflammatory Gene Expressions in Liver Transplant Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Inonu University (Other)
Collaborators: Anadolu University (Other)
Responsible Party: Principal Investigator, Başak KAYHAN, Ph.D. Prof., Prof.Dr., Inonu University
Other Study IDs: 2021/24
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Liver Transplant; Complications; Infections; Gene Amplification; Immune Response
MeSH Terms: conditions — Infections | interventions — Gene Expression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy 13 female 14 male subjects
  Interventions: Genetic: Molecular Immunology , gene expressions
- Transplantation Patients: 10 female, 17 male subjects
  Interventions: Genetic: Molecular Immunology , gene expressions

INTERVENTIONS:
Genetic: Molecular Immunology , gene expressions — Expression levels of inflammatory and anti-inflammatory genes
  Other Names: Diagnostic test

SUMMARY:
In our study, some inflammatory Interleukin-2 , Interleukin-6, Interferon-γ, Tumor Necrosis Factor-α and anti-inflammatory Interleukin-4 and Interleukin-10 cytokine genes expressions and Triggering Receptor Expressed On Myeloid Cells- 1, which contributes to the pathology of acute and chronic inflammatory diseases; Human Leukocyte Antigen-G5, which suppresses the immune response; the expression levels of transcription factor Forkhead box-P3 expressed in regulatory T-lymphocytes and Cluster of Differentiation (CD)14 genes, which are thought to be biomarkers in various infectious diseases and expressed in monocytes, will be measured from peripheral blood samples obtained from liver transplant patients before, 1 month and 6 months after the operation. In addition, the classical liver markers Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Platelet Count (PLT), Alpha Feto Protein (AFP), Direct Bilirubin (Bilirubin D), Total Bilirubin (Bilirubin T) and C- Levels of biochemical parameters such as Reactive Protein (CRP) will be measured. In the light of the data to be obtained, it is aimed to find biomarkers with high predictive value for rejection and infection after liver transplantation.

DETAILED DESCRIPTION:
Liver transplantation is the transplantation of the liver, which is completely or partially removed by surgical intervention, from a living or brain-dead cadaver to the recipient. Today, organ transplantation procedures are carried out successfully in many centers in our country.Liver transplantation has become the most effective treatment method for acute and chronic liver failure due to different reasons.The life expectancy of individuals with advanced liver disease, which was limited to months before liver transplantation, was extended with liver transplantation and the quality of life was improved with this treatment method. However, since most of the organ transplants are made from genetically different donors, tissue compatibility between the donor and the recipient remains a problem.Therefore, the recipient's immune response to donor graft antigens should be considered.

In recent years, the application of advanced surgery and new immunosuppressive approaches has made it possible to successfully transplant almost any vital organ or tissue. However, due to both infection and genetic factors, an immune response to the donor organ may develop and cause organ rejection. At this point, we think that early diagnosis and discovery of immune response parameters that distinguish infection from rejection may be important.In our study, some inflammatory Interleukin-2 , Interleukin-6, Interferon-γ, Tumor Necrosis Factor-α and anti-inflammatory Interleukin-4 and Interleukin-10 cytokine genes expressions and Triggering Receptor Expressed on Myeloid Cells-1, which contributes to the pathology of acute and chronic inflammatory diseases; Human Leukocyte Antigen-G5, which suppresses the immune response; the expression levels of transcription factor Forkhead box-P3 expressed in regulatory T-lymphocytes and Cluster of Differentiation (CD)14 genes, which are thought to be biomarkers in various infectious diseases and expressed in monocytes, will be measured from peripheral blood samples obtained from liver transplant patients before, 1 month and 6 months after the operation. In addition, the classical liver markers Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Platelet Count (PLT), Alpha Feto Protein (AFP), Direct Bilirubin (Bilirubin D), Total Bilirubin (Bilirubin T) and C- Levels of biochemical parameters such as Reactive Protein (CRP) will be measured. In the light of the data to be obtained, it is aimed to find biomarkers with high predictive value for rejection and infection after liver transplantation.

ELIGIBILITY:
Inclusion Criteria: Healthy volunteers without acute or chronic diseases

-

Exclusion Criteria: without acute or chronic bacterial and viral infections; Anti-Hepatitis-C (+), HBsAg (+), Anti-HIV (+), renal failure, neutropenia, using immune supressor medications, autoimmunity (+), acute or chronic pancreatitis, being treated with burns, pregnant, using steroid medications, diabetic patients, any malignancy has been identified and treated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It includes patients who do not disrupt their pre- and post-transplant controls and treatment process, among patients with suitable liver disease, among those whose transplantation decision has been taken in accordance with the protocols of İnönü University Liver Transplantation Institute.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-12-03 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Biochemical parameters | 1st month
  ALT, AST, PLT, AFP, Bilirubin Direct, Bilirubin Total, CRP levels of all subject in control and Transplantation groups before surgery.
Gene expression parameters before surgery | 1st month
  Expression levels of Interleukin-2, Interleukin-6, Interferon-gamma, Tumor Necrosis Factor-alpha, Interleukin-4, Interleukin-10, Triggering Receptors Expressed on Myeloid Cells-1, Human Leukocyte Antigen-G5, Forkhead box p3 and Cluster of Differentiation (CD)14 in peripheral blood samples

SECONDARY OUTCOMES:
Gene Expression parameters after surgery | 2nd-3rd months
  Expression levels of Interleukin-2, Interleukin-6, Interferon-gamma, Tumor Necrosis Factor-alpha, Interleukin-4, Interleukin-10, Triggering Receptors Expressed on Myeloid Cells-1, Human Leukocyte Antigen-G5, Forkhead box p3 and Cluster of Differentiation (CD)14 in peripheral blood samples
Gene Expression parameters after surgery | 4-6th months
  Expression levels of Interleukin-2, Interleukin-6, Interferon-gamma, Tumor Necrosis Factor-alpha, Interleukin-4, Interleukin-10, Triggering Receptors Expressed on Myeloid Cells-1, Human Leukocyte Antigen-G5, Forkhead box p3 and Cluster of Differentiation (CD)14 in peripheral blood samples

OTHER OUTCOMES:
Microbiological analysis | 1st-6th months
  Culture analysis in urine and blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- İnönü University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plans can be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: For 2 years

REFERENCES:
- [Background] Carvalho-Gaspar M, Billing JS, Spriewald BM, Wood KJ. Chemokine gene expression during allograft rejection: comparison of two quantitative PCR techniques. J Immunol Methods. 2005 Jun;301(1-2):41-52. doi: 10.1016/j.jim.2005.03.003. Epub 2005 Apr 1. PMID 16018884
- [Result] Friedman BH, Wolf JH, Wang L, Putt ME, Shaked A, Christie JD, Hancock WW, Olthoff KM. Serum cytokine profiles associated with early allograft dysfunction in patients undergoing liver transplantation. Liver Transpl. 2012 Feb;18(2):166-76. doi: 10.1002/lt.22451. PMID 22006860
- [Result] Hassan L, Bueno P, Ferron-Celma I, Ramia JM, Garrote D, Muffak K, Barrera L, Villar JM, Garcia-Navarro A, Mansilla A, Gomez-Bravo MA, Bernardos A, Ferron JA. Early postoperative response of cytokines in liver transplant recipients. Transplant Proc. 2006 Oct;38(8):2488-91. doi: 10.1016/j.transproceed.2006.08.054. PMID 17097977